CLINICAL TRIAL: NCT04626544
Title: Dynamic Neck Function During Gait in Patients With Dizziness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 169388
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Dizziness; Neck Pain; Gait
MeSH Terms: conditions — Dizziness; Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dizziness: Patients with dizziness referred to a secondary referral center
  Interventions: Device: Body-worn inertial sensors
- Healthy controls: Healthy controls without dizziness or neck pain symptoms for the last 3 months
  Interventions: Device: Body-worn inertial sensors

INTERVENTIONS:
Device: Body-worn inertial sensors — The device typically includes accelerometers that capture body accelerations in three directions (anteroposteriorly, mediolaterally and vertically) and gyrometers that capture rotations (yaw, pitch and roll). The method of measuring gait using body-worn inertial sensors has been found reliable [15] and valid [20]. This project will use Opal sensors and the Mobility Lab software from the manufacturer APDM (https://www.apdm.com/wearable-sensors/).

SUMMARY:
This study aims to explore the possible association between dizziness and head-on trunk-movements and thus, neck movement and if this differs to healthy controls. Additional, the study will examine the reliability and validity of using wearable accelerometers to examine how the head moves relative to the trunk and to collect normative data on head on trunk movement.

DETAILED DESCRIPTION:
Patients with dizziness will be recruited from a ear-nose and throat clinic. After giving written consent the patients will be tested with wearable sensors on their occiput and C6 vertebra during gait. Healthy controls will be recruited from students and employees at the Western Norway University of Applied Science and go through the same protocol as the patients.

The investigators will measure the relationship between the two sensors to explore how patients with dizziness move their-on-trunk during gait.

The projects main hypothesis is that patient with dizziness have reduced attenuation of gait-associated head oscillations with increased coupling of head-on-trunk motion, compared to healthy controls. The neck does not compensate for trunk movements, causing the head to follow the movement of the trunk.

ELIGIBILITY:
Inclusion Criteria:

Locally referred Patients to an ear-nose-and throat (ENT) clinic at an University Hospital for dizziness symptoms.

Exclusion Criteria:

Any severe neurologic or orthopedic disease affecting gait.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with dizziness between the ages of 18 - 70 will be recruited from the ear-nose-and throat (ENT) clinic at Haukeland University Hospital (HUS). The clinic admits approximately 1200 patients yearly referred for dizziness and balance issues. All participants recruited form the ENT-clinic will be examined and diagnosed by an otorhinolaryngologist.
  A group of healthy controls between the ages of 18 - 70 will be recruited to generate normative data. A total of 10 participants of each gender will be recruited in the age groups 18 - 30, 31 - 50, 51 - 70. The participants have to be free of any vestibular symptoms and neck pain, going back the last three months, and they have to be free of any severe neurologic or orthopedic disease affecting gait.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Accelerometer data (anteroposteriorly, mediolaterally and vertically) and gyrometer data (yaw, pitch and roll). | Baseline
  The outcome is the difference/regression between the sensor placed on the participant head and the sensor placed on the participants C6 vertebra. The method of measuring gait using body-worn inertial sensors has been found reliable and valid. This project will use Opal sensors and the Mobility Lab software from the manufacturer APDM (https://www.apdm.com/wearable-sensors/).
Video analysis: Three-dimensional motion capture | Baseline
  Three-dimensional motion capture is considered the gold standard of movement analysis. Using this method, reflective markers are placed on specified body landmarks. The subject is then filmed from different angles using several cameras, allowing for analysis of the markers relative to one another. Both rotation and acceleration is captured this way. The project will use an eight-camera system from Qualisys, with analyses performed using Visual 3D software.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Baseline
  The severity of dizziness handicap will be evaluated using a Norwegian version of the Dizziness Handicap Inventory (DHI) [24]. This questionnaire aims to quantify the handicap experienced by dizziness. It contains 25 items with a maximum score of 100. A score > 29 indicates disability. The Norwegian version of the questionnaire has been validated and the sum score demonstrates satisfactory measurement properties.
Neck Disability Index (NDI) | Baseline
  The degree of neck disability will be measured with the Neck Disability Index (NDI) [26]. The NDI consists of 10 items with each score on a 0 to 5 rating scale and a total range of 0 - 50. Scores between 0-and 4 indicate no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability and 35-50 complete disability [26]. The index has been validated in the evaluation of pain and disability in acute and chronic conditions. The Norwegian version has shown good test-retest reliability.
Vertigo symptom Scale - Short form | Baseline
  To measure the degree of dizziness symptom severity, the Vertigo Symptom Scale - short form (VSSsf) will be used. The form comprise 15 items, and the patients answer how frequently they have experienced symptoms in the past month on a scale from 0-4, giving a range of score from 0 to 60. A higher score indicates increased symptom severity. A score ≥ 12 points on the total scale indicates severe dizziness. The total scale can be subdivided into two subscales measuring severity of autonomic symptoms, such as sweating, heart pounding and nausea, and severity of vertigo and balance symptoms. The questionnaire with its subscales has been validated into Norwegian.
Numeric pain rating scale (NPRS) | Baseline
  Patients reporting neck pain will be asked to rate their neck pain during the two last weeks on an 11-point scale. The NPRS has previously shown adequate reliability and validity in patients with chronic pain conditions, including neck pain.The pain is rated from 0 to 10 where 0 represents no pain and 10 represents the worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Kragerud Goplen, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Høgskulen på Vestlandet, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No